CLINICAL TRIAL: NCT05408767
Title: Accelerated Brain Volume Loss in People With Multiple Sclerosis: do Real-world Observations Align With Standardized Research Findings?
Brief Title: Accelerated Brain Volume Loss in People With Multiple Sclerosis
Acronym: BraVoLoinMS
Status: Completed | Type: Observational
Sponsor: National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Marie D'hooghe, principal investigator, National MS Center Melsbroek
Other Study IDs: BraVoLo in MS
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Retrospective Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore whether brain volume loss (BVL) in people with multiple sclerosis (MS), assessed on magnetic imaging (MRI) data obtained during routine medical follow-up (and thus outside a standardized research environment), differs from that of healthy controls and correlates with measures of physical and/or cognitive disability, the latter also gathered during regular clinical practice.

DETAILED DESCRIPTION:
This project will not be the first study on real-world data in an existing MS cohort. A NMSC research group has already reported on the contribution of a single brain volumetric assessment to the prediction of MS-related disability10 - with distinct patterns for the Expanded Disability Status Scale (EDSS) as a measure of physical disability11, and Symbol Digit Modalities Test (SDMT) as a measure of cognitive disability12 - and found a threshold effect for the lowest brain volumes with regard to SDMT worsening over time10. Ghione and co-workers, in turn, have demonstrated a positive correlation between annualized BVL and EDSS progression based on the EDSS in a very large sample containing nearly 2,000 individuals13. The novelty of this new study lies in the fact that the investigators want to explore the correlations between BVL and changes in an expanded set of routinely collected clinical variables in our center - in addition to the EDSS score - such as Timed 25-Feet Walk Test (T25FWT)14, 9-Hole Peg Test (9HPT)15 and SDMT.

ELIGIBILITY:
Inclusion Criteria:

* MRI and volumetry performed minimum 48 and maximum 60 months apart

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be the difference in annualized whole brain volume percentage change between the MS and control cohort | 4 - 5 years
  the difference in annualized whole brain volume measured by Icometrix

CONTACTS AND LOCATIONS:
Overall Officials: Miguel D'haeseleer, Principal Investigator — National MS center
Locations (1):
- Nationaal Multiple Sclerose Centrum Melsbroek, Melsbroek, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No